CLINICAL TRIAL: NCT05004454
Title: A Randomized, Parallel, Double-blind, Placebo-Controlled Study to Investigate the Effect of a Bacillus Subtilis BS50 Spore Preparation on Gastrointestinal Symptoms in Healthy Adults
Brief Title: Effect of Bacillus Subtilis BS50 Supplementation on Gastrointestinal Symptoms in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIO-CAT Microbials, LLC (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Organization: BIO-CAT, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO-2112
Record Dates: First submitted 2021-07-26; First posted 2021-08-13 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Gastrointestinal Health; Immune Health; Cardiovascular Health; Digestive Health
Keywords: probiotic; Bacillus; subtilis; bloating
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Bacillus subtilis BS50 and placebo powders will be manufactured in to capsules and provided to the clinic in blindly coded containers. The code was generated by parties not responsible for data collection, analysis, or interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacillus subtilis BS50 (Experimental): Subjects will consume 1 capsule containing 2x10⁹ CFU of a Bacillus subtilis BS50 spore preparation once daily for 42 days.
  Interventions: Dietary Supplement: Bacillus subtilis BS50 spore preparation
- Placebo (Placebo Comparator): Subjects will consume 1 capsule containing maltodextrin once daily for 42 days.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis BS50 spore preparation — Subjects will consume 1 capsule containing 2x10⁹ CFU of a Bacillus subtilis BS50 spore preparation once daily for 42 days.
  Arms: Bacillus subtilis BS50
Dietary Supplement: Maltodextrin — Subjects will consume 1 capsule containing maltodextrin once daily for 42 days.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the effect of a novel Bacillus subtilis spore preparation on abdominal bloating, flatulence, and burping in healthy adults.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that, when administered in adequate amounts, confer a health benefit on the host. Examples of probiotic health benefits include the support of gastrointestinal health, immune health, and mood. Common probiotic strains include species from the genera Lactobacillus, Bifidobacterium, and Bacillus. Bacillus species are particularly well suited for probiotic applications because they are often manufactured as spores that persist without refrigeration and show survivability in the acidic conditions of the human gut.

BIO-CAT Microbials' proprietary Bacillus subtilis BS50 strain ("BS50") has previously been shown in bacterial culture to secrete digestive enzymes and candidate gut microbiota-modulating molecules which may help support digestion and gastrointestinal health (unpublished data). BS50 also showed robust heat resistance and pH tolerance, which predicts strain survival across the wide pH range of the human gut. The objective of this clinical study is to investigate the effect of BS50 supplementation at 2x10⁹ CFU per day for 42 days on abdominal bloating, flatulence, and burping in healthy adults.

This study will be a randomized, placebo-controlled, parallel design trial consisting of one screening visit (Visit 1) and two study visits (Visits 2 and 3). At Visit 1 (Day -7), subjects will arrive at the clinic in a fasting state. After subjects provide voluntary informed consent, subjects will undergo medical history, prior and current medication/supplement use, and inclusion and exclusion criteria assessments. Additionally, height, body weight, and vital signs will be measured and BMI will be calculated. Blood samples will be collected for chemistry and hematology analyses. Subjects will also be dispensed a paper Bowel Habits Diary with Bristol Stool Scale (BHD-BSS) and paper Gastrointestinal Tolerance Questionnaire (GITQ) with instructions to capture events occurring during the 7 continuous days prior to Visit 2 (Day 0). The GITQ contains a series of questions regarding the presence and severity of GI symptoms occurring during the past 24 h.

At Visit 2 (Day 0), subjects will arrive at the clinic in a fasting state. Subjects will undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, body weight and vital signs measurements), and adverse event (AE) assessment. The paper BHD-BSS and GITQ will be collected and reviewed. To assess sleep quality and determine presence and duration of respiratory infection, subjects will be instructed to complete a paper Sleep Quality and Respiratory Infection Questionnaire (SQ-RIQ) in the clinic. Blood samples will be collected for assessment of markers of intestinal permeability, inflammation, and lipid profile. Subjects will be randomly assigned to a study product. Subjects will be dispensed their assigned study product and will be instructed to consume it once a day (1 capsule/d) for 42 days starting on Day 0. To assess sleep quality and determine presence and duration of respiratory infection, subjects will be dispensed a weekly electronic SQ-RIQ with instructions to complete this questionnaire weekly prior to Visit 3 (Day 42). Subjects will be dispensed the electronic BHD-BSS and electronic GITQ with instructions to capture events occurring daily leading up to Visit 3 (Day 42).

At Visit 3 (Day 42), subjects will arrive at the clinic fasted and undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, body weight and vital signs measurements), and adverse event (AE) assessment. Blood samples will be collected for chemistry and hematology analyses as well as for assessment of markers of intestinal permeability, inflammation, and lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 30-65 years of age, inclusive at Visit 1.
* BMI of 18.0 to 31.9 kg/m², inclusive, at Visit 1.
* Have ≥3 weekly total symptom score obtained by combining ratings for abdominal bloating, flatulence, and burping from the GITQ.
* Consumes a typical American diet.

Exclusion Criteria:

* Abnormal laboratory test results of clinical significance at Visit 1.
* Clinically important GI condition that would potentially interfere with the evaluation of the study product.
* Recent (within 2 weeks of Visit 1) history of an episode of acute GI illness such as nausea/vomiting or diarrhea.
* Self-reported history (within 6 weeks of Visit 1) of constipation or diarrhea.
* Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders.
* Uncontrolled hypertension as defined by the blood pressure measured at Visit 1.
* Have received a COVID vaccine within 2 weeks of Visit 2 or expected to receive a COVID vaccine during the study period.
* Had a positive SARS-CoV-2 test and experienced symptoms for >2 months.
* History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Weight loss or gain >4.5 kg in the 3 months prior to Visit 1.
* Antibiotic use within 3 months of Visit 1 and throughout the study period.
* Use of steroids within 1 month of Visit 1 and throughout the study period.
* Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDS) within 1 month of Visit 1.
* Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Abdominal bloating, flatulence, and/or burping | 6 weeks
  Daily, 8-item Gastrointestinal Tolerance Questionnaire

SECONDARY OUTCOMES:
Composite score of GI symptoms | 6 weeks
  Abdominal bloating, flatulence, burping, nausea, vomiting, abdominal cramping, stomach rumbling, and reflux (Gastrointestinal Tolerance Questionnaire)
Individual GI symptoms scores other than abdominal bloating, flatulence, and burping | 6 weeks
  Nausea, vomiting, abdominal cramping, stomach rumbling, and reflux (Gastrointestinal Tolerance Questionnaire)
Bowel function | 6 weeks
  Stool frequency, stool consistency, straining and discomfort during bowel movement, sensation of incomplete evacuation (Bowel Habits Diary with Bristol Stool Scale)
Biomarkers of gut permeability | 6 weeks
  Blood levels of zonulin, occludin, and lipopolysaccharide binding protein
Biomarkers of immune health | 6 weeks
  Blood levels of C-reactive protein, IL-8, IL-6, IL-10, IFN-γ, and TNF-α
Blood lipid profiling | 6 weeks
  Blood levels of triglyceride, total cholesterol (total-C), LDL-C, and HDL-C
Incidence and duration of cold/flu/respiratory infection | 6 weeks
  Weekly Sleep Quality and Respiratory Infection Questionnaire
Sleep quality | 6 weeks
  Weekly Sleep Quality and Respiratory Infection Questionnaire
Safety - Adverse Events | 7 weeks
  Self-reported adverse events at Visits 2 and 3
Safety - Blood Chemistry Profile | 7 weeks
  Albumin, alkaline phosphatase, total bilirubin, calcium, chloride, creatinine, blood urea nitrogen, potassium, aspartate, aminotransferase, alanine aminotransferase, sodium, total protein, carbon dioxide, osmolality, and glucose
Safety - Blood Hematology Profile | 7 weeks
  White blood cell count, red blood cell count, hemoglobin concentration, hematocrit (as volume percent), mean cell volume, mean cell hemoglobin, mean cell hemoglobin concentration, neutrophils, lymphocytes, monocytes, eosinophils, basophils, and platelet counts

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (1):
- Biofortis, Merieux Nutrisciences, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garvey SM, Mah E, Blonquist TM, Kaden VN, Spears JL. The probiotic Bacillus subtilis BS50 decreases gastrointestinal symptoms in healthy adults: a randomized, double-blind, placebo-controlled trial. Gut Microbes. 2022 Jan-Dec;14(1):2122668. doi: 10.1080/19490976.2022.2122668. PMID 36269141